CLINICAL TRIAL: NCT01437579
Title: Randomized Controlled Trial for Efficacy of Botulinum Toxin Type A in Treatment of Patients Suffering Bladder Pain Syndrome/Interstitial Cystitis With Hunners' Lesions
Brief Title: Efficacy of Botulinum Toxin Type A in Patients With Bladder Pain Syndrome/Intersticial Cystitis and Hunners' Lesions
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Moscow State University of Medicine and Dentistry (Other)
Responsible Party: Principal Investigator, George Kasyan, Assistant Professor, Moscow State University of Medicine and Dentistry
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BPS/IC Bot1
Record Dates: First submitted 2011-09-18; First posted 2011-09-21 (Estimated); Last update posted 2011-09-21 (Estimated); Status verified 2011-09

CONDITIONS: Interstitial Cystitis
Keywords: interstitial cystitis; bladder pain syndrome; intratrigonal injection; botulinum toxin
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Cystoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulinum toxin (Active Comparator): Bladder intratrigonal injection of botulinum toxin (100 units) in 10 injection sites during cystoscopy under general anesthesia
  Interventions: Procedure: intratrigonal injection of botulinum toxin
- cystoscopy with hydrodistension (Sham Comparator): cystoscopy with hydrodistension under general anesthesia
  Interventions: Procedure: cystoscopy

INTERVENTIONS:
Procedure: intratrigonal injection of botulinum toxin — Bladder intratrigonal injection of botulinum toxin during cystoscopy under general anesthesia
  Arms: Botulinum toxin
Procedure: cystoscopy — cystoscopy under general anesthesia
  Arms: cystoscopy with hydrodistension

SUMMARY:
The etiology of bladder pain syndrome is unknown. Therefore the management is directed to pain relief, as bladder pain is believed to drive both voiding frequency and nocturia. Botulinum toxin A has been shown to decrease noxious input. Several studies showed efficacy of botox for treatment of painful bladder.

The aim of this study is to evaluate the efficacy of Botulinum toxin in patients who are suffering bladder pain syndrome with Hunner lesions during cystoscopy.

ELIGIBILITY:
Inclusion Criteria:

* longer than 6 months of bladder pain syndrome/interstitial cystitis with Hunner Lesion(s) during cystoscopy

Exclusion Criteria:

* Pregnancy
* neurologic diseases
* urinary tract infections
* bladder outlet obstruction
* previous pelvic radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-06; Primary Completion 2011-12 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in pain intensity | 1 week followed by 1, 3, and 6 months after BoNTA injection
  Pain intensity is scored using a 10-point visual analog scale and change from baseline is observed
Change from baseline of intensity of bladder bother symptoms | within 1 week, at 3 months and 6 months
  O'Leary-Sant score was used to assess symptoms and problems.
Change from baseline of quality of life | within 1 week, at 3 months and 6 months
  Quality of life (QoL) was evaluated using question 8 of the International Prostate Symptoms Score.

SECONDARY OUTCOMES:
Postvoid residual urine volume | within 1 week, at 3months and 6 months after BoNTA injection
  uroflowmetry with residual urine measurement
Upper urinary tract retention | 1 week, 3 months and 6 months after BoNTA injection
  Kidney ultrasound investigation

CONTACTS AND LOCATIONS:
Locations (1):
- Urology department of moscow state university of medicine and dentistry, Moscow, Russia

REFERENCES:
- [Derived] Imamura M, Scott NW, Wallace SA, Ogah JA, Ford AA, Dubos YA, Brazzelli M. Interventions for treating people with symptoms of bladder pain syndrome: a network meta-analysis. Cochrane Database Syst Rev. 2020 Jul 30;7(7):CD013325. doi: 10.1002/14651858.CD013325.pub2. PMID 32734597